CLINICAL TRIAL: NCT02117115
Title: Early Post-transplant Contrast-enhanced Abdominal CT to Predict the Risk of Acute Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Abdominal CT to Predict the Risk of Acute Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: GVHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201404063
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic; Multiple Myeloma
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma | interventions — Contrast Media; ioversol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT scan with contrast (Experimental)
  Interventions: Radiation: Dynamic contrast-enhanced computed tomography; Drug: Ioversol

INTERVENTIONS:
Radiation: Dynamic contrast-enhanced computed tomography — CT scan performed between Day +7 and Day +14.
  Other Names: CT scan with contrast
Drug: Ioversol — To optimize visualization of bowel mucosal, patient will be given 1350 ml, or as much as can be tolerated, of negative oral contrast to distend the small bowel one hour prior to scanning. A weight-based volume of Optiray-350 will be injected at a rate of 4 cc/sec followed by 50 cc of saline flush also at 4 cc/sec.
  Other Names: Optiray-350

SUMMARY:
Contrast-enhanced abdominal CT will be performed 1-2 weeks after allogeneic stem cell transplant, and radiographic evidence of mucosal inflammation will be correlated with the subsequent development of acute graft versus host disease. The primary endpoint is the feasibility and safety of contrast-enhanced abdominal CT in the early post-transplant period, as defined by the risk of contrast-related nephropathy or allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of a hematologic malignancy
* Scheduled to undergo allogeneic SCT from a matched sibling donor or an unrelated donor who is 10/10 or 9/10 HLA match. Transplant eligibility is per standard and institutional criteria.
* Age 18-60 years
* Willing and able to provide informed consent

Exclusion Criteria:

* Documented or reported contrast allergy
* Estimated glomerular filtration rate (GFR) < 60
* Deemed too sick by clinician to leave the floor for imaging
* "Nothing-per-mouth" status for other clinical reasons

Inclusion of Women and Minorities

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast related nephropathy | Baseline through 72 hours after intravenous contrast administration
  Contrast related nephropathy is defined as >25% increase in serum creatinine from baseline (day of CT) or 0.5 mg/dL increase in absolute value, within 48-72 hours of intravenous contrast administration.
  Assessed using the National Cancer Institute Common Criteria for Adverse Events (NCI CTCAE) Version 4.0.
  The proportion of patients who develop contrast nephropathy will be recorded.
Incidence of contrast allergic reaction | Within 4 hours after contrast administration
  Assessed using the National Cancer Institute Common Criteria for Adverse Events (NCI CTCAE) Version 4.0.
  The proportion of patients who an allergic reaction will be recorded.

SECONDARY OUTCOMES:
Correlation between CT risk scores and occurrence of acute GVHD | 180 days
  Images will be reviewed for presence of abnormal mucosal enhancement along the gastrointestinal tract including gallbladder and biliary system, bowel wall thickening, engorgement of vasa recta, mesenteric edema, mesenteric lymphadenopathy, bowel wall thickening, and periportal edema. Abnormal GI mucosal enhancement, if present, will be characterized by relative intensity (mild, moderate, severe), number of involved segments (single segment, two segments, or three segments or more), and location of involved segments. Other findings listed above will provide binary data. All data points will then be used for patient risk stratification for developing GvHD.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu